CLINICAL TRIAL: NCT00423852
Title: Phase I/II Trial of Sequential Paclitaxel/Ifosfamide Followed by Dose-Escalated, Dose-Intensive Carboplatin, Paclitaxel and Ifosfamide With Stem Cell Support in Cisplatin-Resistant Germ Cell Tumor Patients
Brief Title: Paclitaxel, Ifosfamide, and Carboplatin Followed By Autologous Stem Cell Transplant in Treating Patients With Germ Cell Tumors That Did Not Respond to Cisplatin
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-077; MSKCC-06077
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Brain and Central Nervous System Tumors; Extragonadal Germ Cell Tumor; Ovarian Cancer; Teratoma; Testicular Germ Cell Tumor
Keywords: recurrent ovarian germ cell tumor; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; recurrent malignant testicular germ cell tumor; adult central nervous system germ cell tumor; stage III malignant testicular germ cell tumor; stage II malignant testicular germ cell tumor; recurrent extragonadal non-seminomatous germ cell tumor; recurrent extragonadal seminoma; stage III extragonadal non-seminomatous germ cell tumor; stage III extragonadal seminoma; stage IV extragonadal non-seminomatous germ cell tumor; stage IV extragonadal seminoma; recurrent extragonadal germ cell tumor; adult teratoma; testicular immature teratoma; testicular mature teratoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Ovarian Neoplasms; Teratoma; Testicular Germ Cell Tumor; Testicular Neoplasms | interventions — Filgrastim; Carboplatin; Ifosfamide; Paclitaxel; Peripheral Blood Stem Cell Transplantation

ARMS (1):
- chemotherapy with Stem Cell Support (Experimental): This is a phase I/II trial of sequential accelerated chemotherapy cycles with paclitaxel/ifosfamide and paclitaxel/ifosfamide and carboplatin administered with G-CSF and PBSC support. During phase I, carboplatin, ifosfamide, and paclitaxel will be dose escalated to determine the MTD. Additional patients will be enrolled in the Phase II portion of the study following the determination of the MTD of Ifosfamide and paclitaxel, to bring the total possible number of patients treated at the MTD to 38.
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: ifosfamide; Drug: paclitaxel; Procedure: autologous hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: ifosfamide
Drug: paclitaxel
Procedure: autologous hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, ifosfamide, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. An autologous peripheral stem cell transplant may be able to replace blood-forming cells that were destroyed by chemotherapy. This may allow more chemotherapy to be given so that more tumor cells are killed.

PURPOSE: This phase I/II trial is studying the side effects and best dose of ifosfamide when given together with paclitaxel and carboplatin followed by an autologous stem cell transplant and to see how well they work in treating patients with germ cell tumors that did not respond to cisplatin.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of paclitaxel and ifosfamide followed by dose-escalated, dose-intensive paclitaxel, carboplatin, and ifosfamide with autologous peripheral blood stem cell support in patients with cisplatin-resistant germ cell tumor. (Phase I)
* Determine the maximum tolerated dose of paclitaxel, carboplatin, and ifosfamide when given with a high-dose treatment program in these patients. (Phase I)
* Determine the efficacy of this regimen when given as salvage therapy in the second-line or third-line setting, in terms of complete response, in these patients. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of paclitaxel, carboplatin, and ifosfamide followed by a phase II, open-label study.

* Phase I:

  * Paclitaxel, ifosfamide, and autologous peripheral blood stem cell (PBSC) collection: Patients receive paclitaxel IV over 3 hours on day 1 and ifosfamide IV over 2 hours on days 1-3. Patients undergo leukapheresis on days 11-13. Patients also receive filgrastim (G-CSF) subcutaneously (SC) twice daily beginning on day 3 and continuing until leukapheresis is completed. Beginning on day 14 or 21, patients may receive a second course of paclitaxel, ifosfamide, and G-CSF. Patients may also undergo additional leukapheresis.
  * Paclitaxel, carboplatin, ifosfamide, and autologous PBSC transplantation: Patients receive paclitaxel IV over 3 hours, high-dose carboplatin IV over 30 minutes, and ifosfamide IV over 4 hours on days 1-3. Patients also receive G-CSF SC beginning on day 3 and continuing until blood counts recover. Patients undergo reinfusion of autologous PBSCs on day 5. Treatment repeats every 21-28 days for 3 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of paclitaxel, carboplatin, and ifosfamide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive treatment as in phase I with paclitaxel, carboplatin, and ifosfamide at the MTD determined in phase I.

After completion of study treatment, patients are followed periodically for 1 year and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed germ cell tumor (GCT)

  * Primary CNS GCT allowed
* Unidimensionally measurable disease OR elevated serum tumor markers (alpha-fetoprotein and/or human chorionic gonadotropin)
* Advanced disease

  * Disease resistant to a cisplatin-based chemotherapy regimen (i.e., failed to achieve a durable complete response to cisplatin)
* Known residual disease after post-chemotherapy surgery allowed

PATIENT CHARACTERISTICS:

* Platelet count ≥ 100,000/mm^3
* WBC ≥ 3,000/mm^3
* Creatinine clearance > 50 mL/min (unless due to tumor obstructing the ureters)
* AST and ALT < 2 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection
* Negative serology for HIV type I and II, human T-lymphotropic virus type I and II, hepatitis B or C virus, syphilis, and cytomegalovirus

  * Hepatitis C negative serology by RIBA or PCR
* Adequate medical condition for general anesthesia

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from recent surgery
* At least 3 weeks since prior chemotherapy
* No prior high-dose therapy with autologous bone marrow transplantation
* No other concurrent chemotherapy
* No other concurrent treatment (e.g., surgery or radiotherapy)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darren Feldman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy With Stem Cell Support: This is a phase I/II trial of sequential accelerated chemotherapy cycles with paclitaxel/ifosfamide and paclitaxel/ifosfamide and carboplatin administered with G-CSF and PBSC support. During phase I, carboplatin, ifosfamide, and paclitaxel will be dose escalated to determine the MTD. Additional patients will be enrolled in the Phase II portion of the study following the determination of the MTD of Ifosfamide and paclitaxel, to bring the total possible number of patients treated at the MTD to 38.
  filgrastim
  carboplatin
  ifosfamide
  paclitaxel
  autologous hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
Period: Overall Study
Arm/Group | Chemotherapy With Stem Cell Support
Started | 26
Completed | 23
Not Completed | 3
Not completed — Removed pior to the high-dose portion | 3

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy With Stem Cell Support
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Response
Description: Response assessed at the completion of therapy (after four to five cycles of chemotherapy and after surgery if necessary)
  Complete Response (CR): A complete response is defined as one of the following:
  * Complete disappearance of all clinical and radiographic and biochemical (normal AFP and HCG) evidence of disease for a minimum of 4 weeks (CR to chemotherapy).
  * Complete disappearance of all biochemical evidence of disease with resection of residual radiographic masses that prove to be negative for residual GCT; this includes both mature teratoma and necrotic debris (CR to chemotherapy) for a minimum of 4 weeks.
  * Complete disappearance of all biochemical evidence of disease with complete surgical excision of all residual radiographic masses that, if pathologically positive for residual malignant GCT, show margins to microscopically free of disease (CR to chemotherapy + surgery). Patients must be free of disease for a minimum of 4 weeks.
Time Frame: 2 year
Measure: Number; unit: participants
Arm/Group | Chemotherapy With Stem Cell Support
Number analyzed (Participants) | 23
participants
  Complete Response (CR) | 12
  Incomplete Response (IR) | 6
  Partial Response (PR) | 5

2. Primary Outcome: Maximum Tolerated Dose of Ifosfamide
Time Frame: 4 years
Measure: Number; unit: mg/m2
Arm/Group | Chemotherapy With Stem Cell Support
Number analyzed (Participants) | 23
mg/m2 | 9990

ADVERSE EVENTS:
Arm/Group | Chemotherapy With Stem Cell Support
Serious Adverse Events (participants affected / at risk) | 9/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy With Stem Cell Support (N=26)
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Febrile neutropenia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Infection w/ Gr 3/4 neut, Blood (Infections and infestations) | 1 (1)
Inf norm ANC/gr1/2 neut-Catheter-related (Infections and infestations) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis/thrombus/embolism (Blood and lymphatic system disorders) | 1 (1)
Edema: head and neck (Blood and lymphatic system disorders) | 1 (1)
Allerg react/hypersens (incl drug fever) (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy With Stem Cell Support (N=26)
ALT, SGPT (Metabolism and nutrition disorders) | 19 (63)
AST, SGOT (Metabolism and nutrition disorders) | 11 (24)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (2)
Alkaline phosphatase (Metabolism and nutrition disorders) | 3 (3)
Amylase (Metabolism and nutrition disorders) | 2 (5)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 9 (14)
Constipation (Gastrointestinal disorders) | 2 (2)
Creatinine (Metabolism and nutrition disorders) | 9 (35)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 12 (20)
Febrile neutropenia (Infections and infestations) | 7 (10)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 23 (115)
Hemoglobin (Metabolism and nutrition disorders) | 25 (100)
Hypotension (Cardiac disorders) | 5 (6)
Infection, other (Infections and infestations) | 2 (2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 25 (100)
Lymphopenia (Blood and lymphatic system disorders) | 26 (100)
Magnesium, high (hypermagnesemia) (Metabolism and nutrition disorders) | 2 (2)
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 18 (45)
Mucositis (Clin exam)- Oral cavity (Gastrointestinal disorders) | 2 (2)
Mucositis (func/sympt)- Oral cavity (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (6)
Neuropathy: sensory (Nervous system disorders) | 7 (12)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 23 (100)
PTT (Blood and lymphatic system disorders) | 3 (5)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 24 (100)
Platelets (Blood and lymphatic system disorders) | 25 (100)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 3 (4)
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 12 (75)
Renal failure (Renal and urinary disorders) | 2 (2)
Sodium, high (hypernatremia) (Metabolism and nutrition disorders) | 2 (7)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 8 (10)
Tinnitus (Ear and labyrinth disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 5 (5)
Lipase (Metabolism and nutrition disorders) | 4 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes